CLINICAL TRIAL: NCT04107597
Title: Myofascial Trigger Point Release and Paced Breathing Training for Chronic Low Back Pain: A Randomized Controlled Trial
Brief Title: Myofascial Trigger Point Release and Paced Breathing Training for Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ARCIM Institute Academic Research in Complementary and Integrative Medicine (Other)
Collaborators: Center für Integrative Therapie Christopher Gordon (Unknown); University Hospital Tuebingen (Other); Die Filderklinik (Unknown); Orthopädisch-Unfallchirurgische Praxis Dr Lembeck & Dr Pampel (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LBP_02
Record Dates: First submitted 2019-09-23; First posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Chronic Low-back Pain
Keywords: Chronic Low-back Pain; Myofascial Trigger Point Release; Core Stabilization Exercises; Paced Breathing Training; Pain Severity; Anxiety; Heart Rate Variability
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Core stabilization exercises (Experimental): Patients with CLBP who practice core stabilization exercises
  Interventions: Other: Core stabilization exercises
- Core stabilization exercises and paced breathing training (Experimental): Patients with CLBP who practice core stabilization exercises combined with paced breathing training
  Interventions: Other: Core stabilization exercises and paced breathing training
- Myofascial trigger point release (Experimental): Patients with CLBP who receive myofascial trigger point release therapy
  Interventions: Other: Myofascial trigger point release
- Myofascial trigger point release and paced breathing training (Experimental): Patients with CLBP who receive myofascial trigger point release therapy combined with paced breathing training
  Interventions: Other: Myofascial trigger point release and paced breathing training

INTERVENTIONS:
Other: Core stabilization exercises — Twelve specific exercises following a standard protocol aiming at an intersegmental stabilization of the spine and strengthening and stabilization of specific muscle groups. The exercises are performed under instruction and supervision by a physiotherapist twice per week for 45 minutes
  Arms: Core stabilization exercises
Other: Core stabilization exercises and paced breathing training — Twelve specific exercises following a standard protocol aiming at an intersegmental stabilization of the spine and strengthening and stabilization of specific muscle groups. The exercises are performed under instruction and supervision by a physiotherapist twice per week for 45 minutes. In addition, the participants practice paced breathing training (before and during the CSE sessions as well as 15 minutes twice per day at home) which has a modulating effect on the autonomic nervous system
  Arms: Core stabilization exercises and paced breathing training
Other: Myofascial trigger point release — A standard protocol of 12 myofascial and trigger point release grips followed by so-called roll-down maneuvers and manual rhythmical oscillation, applied to specific muscles and muscle groups. The treatment is applied twice per week for 45 minutes
  Arms: Myofascial trigger point release
Other: Myofascial trigger point release and paced breathing training — A standard protocol of 12 myofascial and trigger point release grips followed by so-called roll-down maneuvers and manual rhythmical oscillation, applied to specific muscles and muscle groups. The treatment is applied twice per week for 45 minutes. In addition, the participants practice paced breathing training (before and during the MTPR sessions as well as 15 minutes twice per day at home) which has a modulating effect on the autonomic nervous system
  Arms: Myofascial trigger point release and paced breathing training

SUMMARY:
A study to explore whether two different treatment approaches, myofascial trigger point release and core stabilization exercises, both with and without additional paced breathing training, can help patients with chronic low back pain (CLBP) and whether one of the two treatments is superior.

DETAILED DESCRIPTION:
This is a randomized controlled trial to evaluate the effect of myofascial trigger point release therapy compared to core stabilization exercises, both with and without additional paced breathing training, on patients with chronic low back pain (CLBP). The main focus is on changes in pain severity, anxiety and depression, heart rate variability, and use of analgesic medication. Outcomes are measured at baseline (pre-intervention), after ten treatments (post-intervention), at three- and at six-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age between 20 and 70 years
* LBP at least once a week during the last three months
* Pain intensity rated at least 4 on an 11-point scale (0=no pain, 10=worst pain imaginable)
* Muscular pain during flexion, extension and lateral flexion

Exclusion Criteria:

* Acute hernia
* Acute local or generalized inflammation
* Neurological disorders such as multiple sclerosis, Parkinson's disease, hemiplegia
* Fibromyalgia
* Radicular symptoms (Lasègue's sign, weakness of foot dorsiflexion muscle, needles or tingling in the legs)
* Paraspinal tumors or metastases
* Cancer under chemo- or radio-surgical treatment or requiring such during the next 12 months
* Leg prostheses
* Rheumatic, cardiovascular or chronic pulmonary condition precluding 45-minute physical therapy (contraindication declared by a physician)
* Severe depression or severe anxiety currently requiring psychotherapy and/or pharmacotherapy
* Suicidal tendencies
* Drug abuse or addiction
* Pregnancy existing or planned during the study period

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2008-04-01 (Actual); Primary Completion 2008-12-18 (Actual); Study Completion 2009-06-12 (Actual)

PRIMARY OUTCOMES:
Post-intervention pain severity | 5 weeks
  Self-reported severity of LBP after ten treatments with the assigned intervention, assessed with the 4-item pain severity score of the Brief Pain Inventory (BPI). The items are rated on an 11-point scale (0=no pain, 10=worst pain imaginable), the score is reported as the mean of the corresponding items.

SECONDARY OUTCOMES:
Pain severity at three-month follow-up | Measured at three-month follow-up
  Self-reported severity of LBP at three-month follow-up, assessed with the 4-item pain severity score of the Brief Pain Inventory (BPI). The items are rated on an 11-point scale (0=no pain, 10=worst pain imaginable), the score is reported as the mean of the corresponding items.
Pain severity at six-month follow-up | Measured at six-month follow-up
  Self-reported severity of LBP at six-month follow-up, assessed with the 4-item pain severity score of the Brief Pain Inventory (BPI). The items are rated on an 11-point scale (0=no pain, 10=worst pain imaginable), the score is reported as the mean of the corresponding items.
Change in pain interference | Measured at baseline (pre-intervention), 5 weeks (post-intervention), three- and six-month follow-up
  Self-reported LBP-related functional impairment, assessed with the 7-item pain interference score of the Brief Pain Inventory (BPI). The items are rated on an 11-point scale (0=no interference, 10=interferes completely), the score is reported as the mean of the corresponding items.
Change in anxiety | Measured at baseline (pre-intervention), 5 weeks (post-intervention), three- and six-month follow-up
  Assessed with the 7-item subscale Anxiety of the self-reporting Hospital Anxiety and Depression Scale. The items are rated on a 4-point scale (0=positive, 3=negative) and added to a score between 0 (insignificant; non-cases) and 21 (severe)
Change in depression | Measured at baseline (pre-intervention), 5 weeks (post-intervention), three- and six-month follow-up
  Assessed with the 7-item subscale Depression of the self-reporting Hospital Anxiety and Depression Scale. The items are rated on a 4-point scale (0=positive, 3=negative) and added to a score between 0 (insignificant; non-cases) and 21 (severe)
Change in patients' belief in therapists' expertise | Measured at baseline (pre-intervention) and 5 weeks (post-intervention)
  Assessed with the 6-item subscale "Patients' Belief in Therapists' Expertise" of the Questionnaire for Measuring Common Factors in Psychotherapy ("Fragebogen zur Erfassung relevanter Therapiebedingungen", FERT). The items are rated on a seven-point Likert scale (1=totally disagree, 7=totally agree; score between 6 and 42).
Change in patients' expectation of improvement | Measured at baseline (pre-intervention) and 5 weeks (post-intervention)
  Assessed with the 3-item subscale "Patients' Expectation of Improvement" of the Questionnaire for Measuring Common Factors in Psychotherapy ("Fragebogen zur Erfassung relevanter Therapiebedingungen", FERT). The items are rated on a seven-point Likert scale (1=totally disagree, 7=totally agree; score between 3 and 21).
Change in therapists' expectation of improvement | Measured at baseline (pre-intervention) and 5 weeks (post-intervention)
  Assessed with the 3-item scale "Therapists' Expectation of Improvement". The items are rated on a seven-point Likert scale (1=totally disagree, 7=totally agree; score between 3 and 21).
HRV analysis: Change in LF/HF ratio | 24-hour ECG measurements taken at baseline (pre-intervention), 5 weeks (post-intervention), three- and six-month follow-up
  LF/HF ratio = ratio of two bands from frequency domain analysis: LF band (0.04-0.15 Hz), HF band (0.15-0.40 Hz). HRV data are obtained from 24-hour ECG measurements
HRV analysis: Change in SDNN | 24-hour ECG measurements taken at baseline (pre-intervention), 5 weeks (post-intervention), three- and six-month follow-up
  Standard deviation of normal to normal (NN) intervals (ms). HRV data are obtained from 24-hour ECG measurements
HRV analysis: Change in RMSSD | 24-hour ECG measurements taken at baseline (pre-intervention), 5 weeks (post-intervention), three- and six-month follow-up
  Root mean square of successive differences (ms). HRV data are obtained from 24-hour ECG measurements
Change in the use of analgesic medication | Assessed at baseline (pre-intervention), 5 weeks (post-intervention), three- and six-month follow-up
  Amount of analgesic medication according to the medication records kept by the participants

CONTACTS AND LOCATIONS:
Overall Officials: Jan Vagedes, Dr., Principal Investigator — Arcim Institute
Locations (1):
- Arcim Institute, Filderstadt, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be made available, in addition to study protocol and informed consent form.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be made available upon publication for a duration of three months.
Access Criteria: The data will be made available to researchers who provide a methodologically sound proposal for use in achieving the goals of the approved proposal.